CLINICAL TRIAL: NCT05594667
Title: Evaluating the Effect of Length of Time on Selective Serotonin Reuptake Inhibitors (SSRIs) on the Response to Psilocybin-assisted Therapy in Individuals With Mild-moderate Major Depressive Disorder (MDD)
Brief Title: Effect of SSRIs on Response to Psilocybin Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Cybin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cybin-001-Depression
Record Dates: First submitted 2022-10-19; First posted 2022-10-26 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Depression; Major Depressive Disorder; Mild Depression; Moderate Depression; Depressive Disorder
Keywords: Psilocybin
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEX010 (Experimental): 25mg of PEX010 (one-time administration)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 25mg of psilocybin provided by Filament Health
  Other Names: PEX010

SUMMARY:
This study is an open-label, single-arm, within-subjects design in individuals with mild-moderate Major Depressive Disorder (MDD). All participants will receive a single dose of 25mg of psilocybin in a therapeutic setting. In order to investigate the effects of length of time on SSRI therapy, 30 participants with varying lengths of time on SSRI therapy will be enrolled, stratified into four groups:

* Group 1: ≤ 1 year
* Group 2: 1 to ≤ 5 years
* Group 3: 5 to ≤ 10 years
* Group 4: > 10 years

DETAILED DESCRIPTION:
The majority of clinical investigations with psilocybin to date either exclude participants on SSRIs or taper them off SSRIs prior to psilocybin administration. While evidence derived from the use of larger doses of psilocybin suggests that its predominately serotonergic effects are safe when administered in controlled settings, research investigating the effects of psilocybin with individuals taking SSRIs is lacking, despite the prevalent and chronic use of SSRIs in individuals with depression.

The aim of this study is to investigate the effect of length of time on SSRIs on psilocybin-assisted therapy response in individuals with MDD. Specifically, this feasibility study investigates participants who undergo a single-dose of psilocybin (25mg) in combination with pre- and post-dose therapy sessions. The follow-up period in the present study is 12 weeks (3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 19 to 65 years of age
2. Fluent in English
3. Currently receiving treatment with an SSRI (consistent dose for at least 6 weeks), with no changes anticipated throughout the duration of the study
4. QIDS-SR-16 score ≥6
5. Clinically diagnosed Major Depressive Disorder by a psychiatrist prior to screening 5a. Diagnosis defined as meeting the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) criteria (American Psychiatric Association, 2013) for MDD
6. MADRS score 7-34 inclusive (mild-moderate)
7. Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
8. Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study.
9. Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of the drug session day. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
10. Agree that for one week before the drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement (specifically SAM-e, 5-HTP, L-tryptophan, St John's Wort) except when approved by the study Investigator. Exceptions will be evaluated by the Investigator and may include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
11. Agree to refrain from consuming alcohol within two days prior to drug administration.
12. Agree not to take any "as needed" medications on the morning of the drug session.
13. Agree to use of highly effective methods of contraception during the study (females)
14. Normal body mass index (BMI 18.5-24.9)
15. Own an Android or iOS device compatible with the fitness tracker software (Apple iOS 13 or higher, Android OS 7.0 or higher)
16. Able to have a friend or family member pick them up after the dosing session
17. Estimated glomerular filtration rate (eGFR) above 40 mL/min/1.73m2 and all other blood-work values Within Normal Limits

Exclusion Criteria:

1. Current or past history of schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), bipolar disorder, delusional disorder, dissociative disorder, paranoid personality disorder, schizoaffective disorder, borderline personality disorder, anorexia nervosa, bulimia nervosa or substance abuse, as assessed by medical history
2. Currently diagnosed psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain, as assessed by medical history.
3. History of seizures
4. Uncontrolled diabetes, insulin-dependent diabetes, or history of hypoglycemia on oral hypoglycemic agent(s)
5. Paraneoplastic syndrome
6. History of traumatic brain injury within the last 2 years
7. Significantly intrusive PTSD as determined by the Investigator
8. Significant suicide risk as defined by C-SSRS within the past two years
9. Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, vascular or any other major concurrent illness that, in the opinion of the Investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study
10. Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged QTc interval (i.e., QTc > 450msec), artificial heart valve, or TIA in the past year
11. Psychoactive substance use within the previous two months. 11a. The following criteria are preferred: lifetime total psychoactive substance use less than 10 times.
12. Pregnant, nursing or breastfeeding women. Females of childbearing potential must be on a highly effective or double barrier method of contraception, or abstinent.
13. Participation in another clinical trial (currently or within the last 30 days)
14. Current use of rifamycins (rifampin, rifabutin, rifapentine), anticonvulsants (carbamazepine, phenytoin, phenobarbital), nevirapine, efavirenz, taxol, dexamethasone); cytochrome P450 Inhibitors - including all HIV protease inhibitors, verapamil, diltiazem, itraconazole, ketoconazole, erythromycin, clarithromycin, azithromycin, and troleandomycin; ergot alkaloids, pimozide, midazolam, triazolam, lovastatin, simvastatin, fentanyl, warfarin, metoprolol, propranolol, buspirone, tramadol, selegiline, sumatriptan.
15. Current use of inhibitors of UGT1A9 and 1A10, monoamine oxidase inhibitors (MAOIs), Tricyclic antidepressants, aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs).
16. Use of steroids within the past two weeks.
17. Resting blood pressure >140 mmHg systolic and >90 mmHg diastolic at screening

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) | Baseline to end of study (week 12)
  The QIDS-SR16 is a 16-item self-reported rating scale designed to assess severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depression.

SECONDARY OUTCOMES:
QIDS-SR-16 response | Baseline to end of study (week 12)
  Defined as a reduction in score of >50%. The QIDS-SR16 is a 16-item self-reported rating scale designed to assess severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depression.
QIDS-SR-16 remission | Baseline to end of study (week 12)
  Defined as a score of ≤5. The QIDS-SR16 is a 16-item self-reported rating scale designed to assess severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depression.
Montgomery and Asberg Depression Rating Scale (MADRS) | Baseline to end of study (week 12)
  A clinician-rated interview to assess the severity of depression. Each item has a severity scale from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60).
Number of adverse-events (AEs) | Baseline to end of study (week 12)
  Number of reported AEs
Number of serious adverse events (SAEs) | Baseline to end of study (week 12)
  Number of reported SAEs
Recruitment rate | 6 months
  Recruitment feasibility will be defined as a minimum recruitment rate of 70% of our target of 30 individuals within 6 months.
Retention | Through study completion, an average of 6 months
  Retention feasibility will be defined as a retention rate of 90% at study completion

OTHER OUTCOMES:
Electroencephalography (EEG) - Response size of select ERPs (N100, P300, N400) | Baseline to end of study (week 12)
  The NeuroCatch® Platform is an objective, rapid neuro-physiological brain function assessment system, licensed by Health Canada as a Class II medical device. The platform provides acquisition, display, analysis, storage, reporting, and management of EEG and event related potential (ERP) information. Response size will be measured as amplitude in microvolts.
Electroencephalography (EEG) - Response timing of select ERPs (N100, P300, N400) | Baseline to end of study (week 12)
  The NeuroCatch® Platform is an objective, rapid neuro-physiological brain function assessment system, licensed by Health Canada as a Class II medical device. The platform provides acquisition, display, analysis, storage, reporting, and management of EEG and event related potential (ERP) information. Response timing will be measured as latency in milliseconds.
Heart rate variability | 1 month (week -2 to week +2)
  Measured by the WHOOP fitness tracker device
Sleep disturbances | 1 month (week -2 to week +2)
  Measured by the WHOOP fitness tracker device
Time in bed | 1 month (week -2 to week +2)
  Measured by the WHOOP fitness tracker device
Respiratory rate | 1 month (week -2 to week +2)
  Measured by the WHOOP fitness tracker device

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Peters, MD, Principal Investigator — Upstream
Locations (1):
- Centre for Neurology Studies x Upstream, Abbotsford, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No